CLINICAL TRIAL: NCT05147064
Title: Minimally Invasive Surgery Versus Conventional Open Interlaminar Decompression in Treatment of Degenerative Lumbar Canal Stenosis
Brief Title: Minimal Invasive Surgery Versus Interlaminar Decompression in Lumbar Canal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Garamoun Abd El Zaher, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Minimal invasive surgery LCS
Record Dates: First submitted 2021-10-22; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Lumbar Spinal Stenosis
Keywords: minimally invasive surgery; interlaminar decompression
MeSH Terms: conditions — Spinal Stenosis | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): randomly allocated
  Interventions: Procedure: minimally invasive surgery
- group B (Experimental): randomly allocated
  Interventions: Procedure: conventional open surgery

INTERVENTIONS:
Procedure: minimally invasive surgery — using (tubular dilators, surgical microscope, and/ or endoscope). the other group will be operated by conventional inter laminar decompression.
  Arms: group A
Procedure: conventional open surgery — open interlaminar lumbar decompression
  Arms: group B

SUMMARY:
Conventional open surgery has been shown to be an effective procedure for LCS decompression. Minimally invasive surgery (MIS) through tubular retractors is a recently introduced alternative procedure for decompression of LCS.

The current study aims at evaluating the efficacy of minimally invasive surgery as a decompressive procedure in comparison to conventional open surgery for the treatment of patients with LCS.

DETAILED DESCRIPTION:
Lumbar canal stenosis (LCS) is defined as narrowing of the spinal canal, the vertebral foramina, and/or the lateral recesses, causing compression on the nearby neurologic structures. Degenerative LCS is one of the most common reasons for old patients to undergo spinal surgery. Neurogenic claudication is the most common symptom for LCS patients. The patients complain of pain or discomfort that radiates to the buttock, thigh and lower limb after walking for a certain distance, therefore leading to functional disability and decreased walking capacity. Conservative management is the first line of treatment in the absence of progressive neurologic deficit or intractable pain, consisting of physical therapy, medications (analgesics, steroids) and pain management procedures. Surgical intervention is recommended if the symptoms are persistent or worsening.

Various techniques are currently used for direct decompression of LCS. Conventional open surgery involves laminectomy that has been shown to be an effective procedure for LCS decompression. However, wide laminectomies disturbs the stability of bony and ligamentous structures and may exacerbate preexisting spondylolisthesis. Minimally invasive surgery (MIS) through tubular retractors is a recently introduced alternative procedure for decompression of LCS. This technique avoids detachment of the paraspinal muscles and may promote preservation of stabilizing ligamentous and bony spinal structures.

The current study aims at evaluating the efficacy of minimally invasive surgery as a decompressive procedure in comparison to conventional open surgery for the treatment of patients with LCS.

ELIGIBILITY:
Inclusion Criteria:

* all patient with lumbar canal stenosis From 18_70 years old

Exclusion Criteria:

* instability Infection Tumours of vertebrae

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | Change of ODI is being assessed immediate pre operatively, after 3, 6,and 12 months post operatively.
  Change of Oswestry disability index (ODI) is being assessed to compare the pre and post operative values.
  This outcome measure is designed to assess function in activities of daily living for those with acute or chronic back pain.
  The ODI consists of 10 patient-completed questions in which the response options are presented as 6-point Likert scales. Scores range from 0% (no disability) to 100% (most severe disability).
back pain and lower limb pain | using visual analogue scale change of the values is being assessed immediate pre operatively, after 3, 6,and 12 months post operatively.
  Change of visual analogue scale (VAS) is being assessed to compare the pre and post operative values. VAS is a continuous scale comprised of a horizontal line, usually 10 centimeters in length. For pain intensity, "no pain" (score of 0) or "worst imaginable pain" (score of 10).

SECONDARY OUTCOMES:
Intraoperative blood loss | intraoperative
  amount of intraoperative blood loss
Operative time | intraoperative
  in minutes